CLINICAL TRIAL: NCT01662037
Title: Bosentan Therapy for High Risk Staged Fontan Procedure in Children With Functional Single Ventricle
Brief Title: Bosentan Therapy in Children With Functional Single Ventricle
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Limin Zhu, Attendant doctor, Department of thoracic and cardiovascular surgery, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJTUMS-20120314
Record Dates: First submitted 2012-08-05; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Congenital Heart Defects; Functional Single Ventricle
Keywords: Pulmonary vascular resistance; Heart defects, Congenital; Receptors, endothelin; Bosentan
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bosentan group (Experimental): Bosentan 2mg/kg/dose twice a day and routinely therapy in children with functional single ventricle during the period of staged Fontan procedure with high risk of increased PVR.
  Interventions: Drug: Bosentan
- Routinely group (No Intervention): Routinely therapy in children with functional single ventricle during the period of staged Fontan procedure with high risk of increased PVR.

INTERVENTIONS:
Drug: Bosentan — Bosentan 2mg/kg/dose twice a day and routinely therapy in children with functional single ventricle during the period of staged Fontan procedure with high risk of increased PVR.
  Other Names: Tracleer
  Arms: Bosentan group

SUMMARY:
Bosentan is a kind of dual endothelin receptor antagonist.The purpose of this study is to investigate if Bosentan therapy can modify the outcome of children with functional single ventricle.

DETAILED DESCRIPTION:
Increased pulmonary vascular resistance (PVR) is a serous issues in children with functional single ventricle during the staged operative period. The purpose of this study is to investigate if Bosentan therapy can improve the survival and life quality after staged Fontan procedure in the children with high risk of increased PVR.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained from patient's legally acceptable representative.
* Pediatric patients waiting for staged Fontan procedure with high risk of increased PVR after bidirectional cavopulmonary connection (BCPC)

  * Transpulmonary pressure gradiant (TPG) > 10mmHg when the obstruction of anastomosis and lung problem were excluded.
  * With the diagnosis of high risk of increased PVR, such as associated with TAPVC, after pulmonary artery banding, after systemic to pulmonary shunt more than 6 months, and et al.
  * Diagnosed as increased PVR with catheterization.

Exclusion Criteria:

* PAH associated with conditions other than those mentioned above, e.g., iPAH, PAH secondary to portal hypertension, HIV patient with opportunistic infection
* Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements
* AST and/or ALT > 3 times the upper limit of normal ranges.
* Hemoglobin concentration < 75% the lower limit of normal ranges
* Treatment or planned treatment with another investigational drug within 3 months of screening
* Treatment with calcineurin-inhibitors (e.g., cyclosporine A and tacrolimus), fluconazole, glibenclamide (glyburide) within 1 week of enrollment of this study
* Known hypersensitivity to bosentan or any of the excipients

Ages: 4 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay and ICU stay | 12 months after Fontan operation

SECONDARY OUTCOMES:
Symptoms of increased PVR | 12 months after Fontan operation
  facial edema plural effusion pericardium effusion
WHO functional class | 12 months after Fontan operation

CONTACTS AND LOCATIONS:
Overall Officials: Zhuoming Xu, MD PhD, Study Director — Cardiac intensive care unit, Department of Thoracic and cardiovascular Surgery, Shanghai children's Medical Center
Locations (1):
- Cardiac intensive care unit, Department of cardiothoracic vascular surgery, Shanghai Children's Medical Center, Medical college of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China